CLINICAL TRIAL: NCT05091788
Title: Clinical Evaluation of the Safety and Efficacy of Aime Robotic Mechanical Coring Device for the Treatment of Moderate to Severe Facial Wrinkles
Brief Title: Robotic Mechanical Coring for the Treatment of Moderate to Severe Facial Wrinkles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI0321
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Wrinkle
Keywords: Wrinkles; Mechanical Coring; Robotic Coring; Skin Coring; Rhytides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Experimental): All subjects will receive two coring treatments on the cheeks with the robotic coring device.
  Interventions: Device: Venus Aime

INTERVENTIONS:
Device: Venus Aime — Venus Aime is a micro-coring device of the skin that can potentially help reduce moderate to severe facial wrinkles.
  Other Names: Aime

SUMMARY:
This study is a prospective, up to 4 center study of the safety and efficacy of mechanical coring with skin closure of cored holes, intended for the improvement in the appearance of wrinkles of the cheeks in up to 70 subjects after two treatments.

DETAILED DESCRIPTION:
Prospective, up to 4 center study of the safety and efficacy of mechanical coring with Tegaderm tape skin closure of cored holes to achieve improvement in the appearance of wrinkles of the cheeks. The study will evaluate the progress of up to 70 subjects after two treatments on the cheeks. Up to 70 subjects who meet inclusion/exclusion criteria will be treated. All subjects will be monitored for a period 7, 37, 60 and 120 days post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between 22 and 75 years of age.
2. Able to read, understand and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Women of childbearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study and have a negative Urine Pregnancy test at baseline.
5. Fitzpatrick skin type I to IV.
6. Cheek areas are at least a score of 3 using the Lemperle Wrinkle Scale as judged by the Investigator.

Exclusion Criteria:

1. Previous aesthetic (device and/or surgical) skin treatment (injection of dermal fillers, fat, or botulinum toxin), in the treated areas in the last 6 months.
2. Silicone, Tattoos, body jewelry, that cannot be removed for the duration of treatment and/or any other synthetic material in the treatment area.
3. Any type of scar in the treatment area
4. Excessive sun exposure and use of tanning beds or tanning creams within 30 days to prior to treatment.
5. History of keloid formation or hypertrophic scarring.
6. Active smoker or having quit smoking in the last 3 months.
7. Active, chronic, or recurrent infection including Herpes simplex virus (HSV) infection or history of HSV in the last 6 months.
8. Compromised immune and/or healing system (e.g., poorly controlled diabetes, collagen vascular disease or autoimmune diseases such as scleroderma, morphea, etc.).
9. Hypersensitivity/allergy to analgesic agents, Betadine, tumescent, Tegaderm or tensioning tape that will be used in the study.
10. Co-morbid condition that could limit the ability of the subject to participate in the study or to comply with follow-up requirements.
11. Pregnant, planning pregnancy during the trial course or breastfeeding.
12. History of bleeding disorder or taking medication that can potentially increase bleeding including anticoagulation.
13. Carcinoma, melanoma, or any other cutaneous cancerous condition in the last 6 months.
14. Non-cancerous lesions (e.g. actinic keratosis, vitiligo, cutaneous papules, nodules, active inflammatory lesions) in the region to be treated.
15. Currently or in the last 1-month part of another clinical study of an investigational drug and/or experimental medical device.
16. Any medical condition that, at the discretion of the investigator, would hamper the impact or the healing process and contra-indicate the subject's participation.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of correct identification of photograph sets from baseline and Day 120 | 4 Months
  Proportion of correct identification of photograph sets from baseline and Day 120 as assessed by independent blinded evaluators. This proportion of correct identification should be greater than completely random theoretical percentage of 0.5. Statistical significance (p<0.05) should be shown using one-sided binomial test comparing to 0.5.

SECONDARY OUTCOMES:
Assess aesthetic improvement using Global Aesthetic Improvement Scale | 4 Months
  Overall aesthetic improvement as assessed using the Global Aesthetic Improvement Scale (GAIS) by the Investigator at Day 120 compared to baseline
  Very much improved (Optimal cosmetic result) = 5, Much Improved (Marked improvement from initial condition, but not completely optimal)=4, Improved (Obvious improvement in appearance from initial condition, but re-treatment is indicated)=3, No Change (The appearance is essentially the same as original condition)=2, Worse (The appearance is worse than the original condition)
Assess subject satisfaction post-treatment using Subject Satisfaction Scale | 4 Months
  Subject satisfaction as assessed using the Subject Satisfaction Scale (SSS) completed by subjects on Day 120. Satisfaction with the aesthetic appearance of the treatment area.
  Very Satisfied=4, Satisfied=3, Having No Opinion=2, Unsatisfied=1, Very Unsatisfied=0

OTHER OUTCOMES:
Assess subject's assessment of discomfort and pain using Visual Analogue Scale | 1 day
  Subjects' assessment of discomfort and pain after treatments as measured using the VAS Pain Scale immediately after treatment
Assess safety profile by recording adverse events | 4 Months
  Subjects experiencing a treatment-related adverse event (AE) in the first 120 days post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, PhD, Study Director — Venus Concept
Locations (2):
- United States (2):
  - DeNova Research, Chicago, Illinois
  - Dermatology, Laser & Vein Specialists of the Carolinas, PLLC, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No